CLINICAL TRIAL: NCT04008381
Title: Efficacy and Safety of Ex-vivo Expanded γδ T Lymphocytes in Patients With Refractory/Relapsed Acute Myeloid Leukaemia: a Single-center, Open-label, Single-arm Clinical Study.
Brief Title: Ex-vivo Expanded γδ T Lymphocytes in Patients With Refractory/Relapsed Acute Myeloid Leukaemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Jinan University, China (Unknown)
Responsible Party: Principal Investigator, MEI HENG, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WHUH-2009-V010
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: gamma-delta T; Refractory/Relapsed
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ex-vivo Expanded γδ T Lymphocytes (Experimental): Patients receive ex-vivo expanded γδ T Lymphocytes (Dose escalation, 2*10^6, 4*10^6, 8*10^6 of cells per kg of body weight).
  Interventions: Biological: Ex-vivo Expanded γδ T Lymphocytes

INTERVENTIONS:
Biological: Ex-vivo Expanded γδ T Lymphocytes — Patients receive ex-vivo expanded γδ T Lymphocytes (Dose escalation, 2*10^6, 4*10^6, 8*10^6 of cells per kg of body weight).

SUMMARY:
This study investigates the potential curative properties of ex-vivo expanded gamma delta T-cells obtained from a blood-related donor for patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm study to evaluate the safety and efficacy of ex-vivo expanded γδ T-lymphocytes in patients with relapsed or refractory acute myeloid leukemia. PBMCs will be separated from peripheral blood of suitable donors. After making them potential cancer killer γδ T Cells, they will be infused to the patients as an immunotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. History of acute myeloid leukaemia (initially diagnosed by presence of 20% or more blast cells with myeloid or monocytic differentiation confirmed by flow cytometry in peripheral blood or bone marrow)
2. Relapsed or refractory AML. A. AML relapse after intensive chemotherapy; B. AML relapse after allogeneic HCT; C. AML progression on low intensity therapy (low dose cytarabine, 5-azacytidine or decitabine); D. No response to at least 4 cycles of low intensity therapy; E. AML refractory to 2 cycles of induction chemotherapy.
3. Presence of > 5% of blasts in bone marrow or peripheral blood smear
4. Patient not eligible for or does not consent to high dose salvage chemotherapy and/or allogeneic Haematopoietic Cell Transplantation (HCT)
5. Considered suitable for lymphodepleting chemotherapy
6. The patient's peripheral superficial venous blood flow smoothly, which can meet the needs of intravenous drip.
7. Patient's main organs function well. A. Liver function: ALT/AST < 3 times the upper limit of normal (ULN); B. total bilirubin≤34.2μmol/L; C. Renal function: Creatinine < 220μmol/L; D. Pulmonary function: Indoor oxygen saturation≥95%; E. Cardiac Function: Left ventricular ejection fraction (LVEF) ≥40%;
8. Life expectancy of at least 3 months
9. Patient ECOG score≤2, Estimated survival time≥3 months.
10. Ability to be off systemic prednisone and other immunosuppressive drugs for at least 3 days prior to γδ T cells product infusion. Maintenance replacement steroid is allowed.
11. The patients did not receive any anticancer treatments such as chemotherapy, radiotherapy and immunotherapy (such as immunosuppressive drugs) within 4 weeks before admission, and the toxicity related to previous treatments had returned to < 1 level at admission (except for low toxicity such as alopecia).
12. Patient able to understand and sign written informed consent
13. Age 18 years up to the age of 75 (≤ 75)

Exclusion Criteria:

1. Women who are pregnant (urine/blood pregnancy test positive) or lactating.
2. Male or female with a conception plan in the past 1 years.
3. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 1 years after enrollment.
4. Uncontrolled infectious disease within 4 weeks prior to enrollment.
5. Active hepatitis B/C virus.
6. HIV infected patients.
7. Suffering from a serious autoimmune disease or immunodeficiency disease.
8. The patient is allergic and is allergic to macromolecular biopharmaceuticals such as antibodies or cytokines.
9. The patient participated in other clinical trials within 6 weeks prior to enrollment.
10. Systemic use of hormones within 4 weeks prior to enrollment (except for patients with inhaled corticosteroids).
11. Have a history of epilepsy or other central nervous system diseases.
12. Having drug abuse/addiction.
13. According to the researcher's judgment, the patient has other unsuitable grouping conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Four-months remission rate | 4 months
  Number of patients reaching Complete Remission (CR) according to National Comprehensive Cancer Network (NCCN, Version 1.2015).
Number of participants with adverse events (AEs) | 3 years
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0).

SECONDARY OUTCOMES:
Overall survival | 3 years
  OS was calculated from the first infusion to death or last follow-up (censored).
Event-free survival | 3 years
  EFS was calculated from the first infusion to death, progression of the disease, relapse or gene recurrence, whichever came first, or last visit (censored).
Relapse-free survival | 3 years
  RFS was calculated from the first infusion to relapse or last visit (censored).
Quantity of gamma-delta T cells in bone marrow cells and peripheral blood cells | 3 years
  Persistence of γδ T cells assessed by number and phenotype of γδ T cells using flow cytometry assay in peripheral blood and bone marrow from patients
lymphocyte subsets function assessment of bone marrow cells and peripheral blood cells | 3 years
  Assessment of lymphocyte subsets function using flow cytometry assay in peripheral blood and bone marrow from patients.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, M.D. Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No